CLINICAL TRIAL: NCT02703220
Title: Pathophysiology-Guided Therapy for Sleep Apnea in the Elderly
Brief Title: Sleep Apnea in Elderly
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PULM-008-14F
Record Dates: First submitted 2016-01-29; First posted 2016-03-09 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea; Elderly Adults
Keywords: sleep apnea; chemoresponsiveness; cerebrovascular response; hyperoxia; acetazolamide; finasteride; apneic threshold; carbon-dioxide reserve
MeSH Terms: conditions — Sleep Apnea Syndromes; Hyperoxia | interventions — Oxygen; Acetazolamide; Finasteride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hyperoxia (Experimental): Determine the effect of sustained hyperoxia overnight vs room air overnight on ventilatory control during sleep, including the apneic threshold, carbon-dioxide reserve and chemosensitivity measured via pressure support ventilation (PSV) during (non-rapid eye movement sleep) NREM sleep.
  Interventions: Other: Hyperoxia/oxygen
- Acetazolamide (ACZ) (Experimental): Determine the effect of acetazolamide on cerebrovascular responsiveness to CO2 during wake and sleep. Participants will receive oral ACZ therapy for 7 days prior to the experimental night, on the night of the study and the subsequent night when polysomnography (PSG) will be performed.
  Interventions: Drug: Acetazolamide
- Finasteride (Experimental): Determine the effect of oral finasteride therapy vs placebo for 1 month on SDB and the AT and chemosensitivity during NREM sleep.
  Interventions: Drug: Finasteride

INTERVENTIONS:
Other: Hyperoxia/oxygen — The ventilatory effects of brief hyperoxia will be assessed by analyzing control breaths on room air immediately preceding the hyperoxic exposure, and comparing with the primary end-point, nadir minute ventilation breath, immediately following the brief hyperoxic exposure
  Arms: Hyperoxia
Drug: Acetazolamide — Participants with sleep apnea will ingest capsules containing either placebo or acetazolamide 500 mg twice a day for 5 days. On the final 2 consecutive nights while still on ACZ, the investigators will perform i) physiology tests and ii) in-lab follow-up PSG.
  Arms: Acetazolamide (ACZ)
Drug: Finasteride — Elderly males with sleep apnea and adequate testosterone levels will ingest placebo vs finasteride, at 5 mg a day for 1 month (mo). After 1 mo, while still on the drug, on the final 2 consecutive nights, the investigators will perform i) physiology tests and ii) in-lab follow-up PSG. Blood tests will be performed to check sex hormone levels. A washout period of 1 month prior to cross-over to the alternate arm (placebo).
  Arms: Finasteride

SUMMARY:
Sleep-disordered breathing (SDB or sleep apnea) is very common among elderly Veterans and leads to increased morbidity and mortality in this population. The proposal aims to identity whether oxygen, finasteride and acetazolamide can be effective in reducing unstable breathing and eliminating sleep apnea in the elderly via different mechanisms. This proposal will enhance the investigators' understanding of the pathways that contribute to the development of sleep apnea in the elderly. The investigators expect that the results obtained from this study will positively impact the health of Veterans by identifying new treatment modalities for sleep apnea. A cumulative effect of the investigators' research will fulfill the long-term goal of improving the quality of life of elderly Veterans suffering from sleep apnea and its potential life-threatening complications.

DETAILED DESCRIPTION:
Sleep apnea-hypopnea syndrome (SAHS) has a high prevalence and is associated with adverse cardiovascular consequences in elderly Veterans. Positive airway pressure therapy is deemed cumbersome and often associated with non-adherence to therapy. This proposal will investigate whether alternative therapies can be developed by modulating specific physiologic mechanisms of ventilatory control. Specifically, the investigators will study whether interventions with sustained hyperoxia (Aim 1), finasteride (Aim 2) and acetazolamide (Aim 3) will reduce breathing instability during sleep by reducing chemoresponsiveness and/or increasing cerebrovascular reactivity (CVR) in order to alleviate sleep disordered breathing in the elderly with sleep apnea. The proposed aims will also allow us to delineate key mechanisms of breathing instability in the elderly. The investigators envision that the results obtained from this project will ultimately allow us to develop novel alternative therapies for sleep apnea in the elderly. We will also compare CVR in young vs older adults

ELIGIBILITY:
Inclusion Criteria:

* Adults who are 60 years old and older, with mild to moderate sleep apnea with AHI >/=5 to 20/hr with central, obstructive, mixed apneas and hypopneas.
* For the finasteride protocol elderly men with above criteria will be enrolled.

Exclusion Criteria:

* Patients with severe sleep apnea (AHI>20/hr)
* Patients with history of prostate cancer
* Males with hypogonadism
* History of cardiac disease, including myocardial infarction
* Bypass surgery
* Atrial and ventricular tachy-bradycardias
* Systolic congestive heart failure and Cheyne-Stokes respiration
* Current unstable angina
* Stroke
* Schizophrenia
* Untreated hypothyroidism
* Seizure disorder
* Preexisting renal failure and liver disorders
* Failure to give informed consent.
* Patients with significant pulmonary diseases by history and abnormal pulmonary function testing, including moderate obstructive/restrictive lung/chest wall disorders with resting oxygen saturation of <96% or on supplemental oxygen
* Patients on certain medications including:

  * study drugs
  * sympathomimetics/parasympathomimetics or their respective blockers
  * narcotics
  * antidepressants
  * anti-psychotic agents
  * other central nervous system (CNS) altering medications
  * current alcohol, tobacco or recreational drug use
* Patients with BMI>34kg/m2 will be excluded to avoid the effects of morbid obesity on pulmonary mechanics and ventilatory control
* Elderly with unstable gait or mobility issues that may preclude safe participation
* Individuals with allergy to finasteride or acetazolamide will be excluded from the specific protocol
* Pregnant women

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The Finasteride arm of the study is only applicable for male gender.
Enrollment: 100 (Estimated)
Dates: Start 2015-07-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Apneic threshold- a measure of breathing instability | 2 days to 30 days
  Measures of breathing instability including: Apneic threshold: this is the end-tidal Co2 at which a central apnea closes to a hypopnea is produced.
Cerebrovascular responsiveness to carbon-dioxide | 7 days
  Cerebrovascular response to different levels of CO2: this is a measure of the response of the cerebral blood flow to changes in carbon dioxide levels and is used as a measure of ventilatory control of breathing
Ventilatory responsiveness | 2 days to 30 days
  Hypocapnic ventilatory response; this is calculated as the change in minute ventilation for corresponding changes in PETCO2.
Carbon -dioxide reserve | 2 days to 30 days
  This is a derived measure. This is calculated as the difference between the apneic threshold PETCO2 (given above) and the control PETCO2.

SECONDARY OUTCOMES:
Apnea hypopnea index | 2 days to 30 days
  Apnea hypopnea index- is a measure of severity of sleep apnea - this is calculated as the total number of apneas and hypopneas recorded during a sleep study divided by the total sleep time during the sleep study.

CONTACTS AND LOCATIONS:
Overall Officials: Susmita Chowdhuri, MD MS, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No